CLINICAL TRIAL: NCT07104383
Title: A Phase 3 Randomized, Double-Blind, Placebo-Controlled, 78-Week Efficacy and Safety Study of VK2735 Administered Subcutaneously for Weight Management in Participants With Type 2 Diabetes Who Are Obese, or Overweight
Brief Title: VK2735 for Weight Management Type 2 Diabetes Phase 3 (VANQUISH 2)
Status: Recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Viking Therapeutics, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: VK2735-302
Record Dates: First submitted 2025-07-29; First posted 2025-08-05 (Actual); Last update posted 2026-02-10 (Actual); Status verified 2026-02

CONDITIONS: Weight Loss
MeSH Terms: conditions — Weight Loss

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (4):
- Placebo Assignment (Placebo Comparator): VK2735 Placebo Comparator Once Weekly
  Interventions: Drug: VK2735
- Active Assignment (Dose #1) (Experimental): VK2735 7.5mg Once Weekly
  Interventions: Drug: VK2735
- Active Assignment (Dose #2) (Experimental): VK2735 12.5mg Once Weekly
  Interventions: Drug: VK2735
- Active Assignment (Dose #3) (Experimental): VK2735 17.5mg Once Weekly
  Interventions: Drug: VK2735

INTERVENTIONS:
Drug: VK2735 — VK2735 is a peptide GLP-1 and GIP dual agonist administered Once Weekly

SUMMARY:
This is a phase 3, multicenter, 78-week randomized, double-blind, placebo-controlled, parallel arm study that will evaluate the weight loss efficacy as well as safety, tolerability, pharmacodynamic effects, and pharmacokinetics of VK2735 in adults with Type 2 Diabetes who are obese or overweight

ELIGIBILITY:
Inclusion Criteria:

1. Age ≥18 years of age at the time of signing the informed consent
2. Body mass index (BMI) ≥27 kg/m2
3. Have Type 2 Diabetes Mellitus according to the American Diabetes Association with HbA1c ≥ 7% to ≤ 11% at screening, on stable therapy for the last 3 months prior to Screening. Type 2 diabetes mellitus may be treated with diet/exercise alone or any oral glycemic-lowering agent (as per local labeling), EXCEPT for amylin analogues or dipeptidyl peptidase 4 (DPP-4) inhibitors or GLP-1R agonists or dual GLP-1/ glucose-dependent insulinotropic polypeptide (GIP) receptor agonists

Exclusion Criteria:

1. History of or current clinically significant medical disorder that, in the opinion of the Investigator, does not support study participation
2. Self-reported body weight change of 5% or more within 3 months of screening
3. Have a prior or planned surgical treatment for obesity (except for liposuction or abdominoplasty if performed >1 year prior to screening)
4. Have or plan to have endoscopic and/or device-based therapy for obesity or have had device removal within the last 6 months prior to screening (such as mucosal ablation, gastric artery embolization, intragastric balloon, duodenal-jejunal endoluminal line)
5. Have Type 1 diabetes mellitus, history of ketoacidosis or hyperosmolar state/coma or any other types of diabetes except Type 2 diabetes mellitus (T2DM)
6. Have had 1 or more episodes of severe hypoglycemia and/or 1 or more episode of hypoglycemia unawareness within 6 months of screening

   • Note: Severe hypoglycemia episodes should be considered when severe cognitive impairment requiring the assistance of another person occurs and the administration of carbohydrate, glucagon, or other resuscitative actions are required. Blood glucose (BG) measurements may not be available during such an event, but neurological recovery attributable to the restoration of BG to normal is considered sufficient evidence that the event was induced by a low BG concentration. If BG measurements are available, the levels associated with severe hypoglycemia are BG < 54 mg/dL
7. Have at least 2 confirmed fasting self-monitoring blood glucose (SMBG) values > 270 mg/dL (on 2 non-consecutive days) within 4 weeks prior to randomization
8. Have proliferative diabetic retinopathy OR diabetic macular edema OR non-proliferative diabetic retinopathy that requires acute treatment
9. Personal or family history of medullary thyroid carcinoma (MTC) or multiple endocrine neoplasia type 2 (MEN2)
10. History of acute or chronic pancreatitis
11. Thyroid disease that is not controlled (Thyroid stimulating hormone (TSH) outside normal range by central lab at screening; one repetition during screening is allowed). Participants with previous history of partial/total thyroidectomy or hypothyroidism may be included, provided their hormone replacement dose has been stable for 3 months prior to screening

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1100 (Estimated)
Dates: Start 2025-06-23 (Actual); Primary Completion 2027-07-01 (Estimated); Study Completion 2027-08-01 (Estimated)

PRIMARY OUTCOMES:
Percent change in body weight from baseline to Week 78 in body weight | 78 Weeks

SECONDARY OUTCOMES:
Percentage of participants who achieve ≥5%, ≥10%, ≥15% and ≥20% body weight reduction after 78 weeks of treatment | 78 Weeks

CONTACTS AND LOCATIONS:
Locations (134):
- United States (132):
  - Viking Clinical Site #2037, Birmingham, Alabama
  - Viking Clinical Site #2064, Birmingham, Alabama
  - Viking Clinical Site #2128, Huntsville, Alabama
  - Viking Clinical Site #2081, Mobile, Alabama
  - Viking Clinical Site #2005, Chandler, Arizona
  - Viking Clinical Site #2017, Flagstaff, Arizona
  - Viking Clinical Site #2018, Peoria, Arizona
  - Viking Clinical Site #2135, Scottsdale, Arizona
  - Viking Clinical Site #2019, Tucson, Arizona
  - Viking Clinical Site #2036, Little Rock, Arkansas
  - Viking Clinical Site #2071, Chula Vista, California
  - Viking Clinical Site #2070, Escondido, California
  - Viking Clinical Site #2054, Huntington Park, California
  - Viking Clinical Site #2014, Lake Forest, California
  - Viking Clinical Site #2129, Lemon Grove, California
  - Viking Clinical Site #2051, Lincoln, California
  - Viking Clinical Site #2050, Long Beach, California
  - Viking Clinical Site #2055, Los Angeles, California
  - Viking Clinical Site #2078, Manteca, California
  - Viking Clinical Site #2053, Montclair, California
  - Viking Clinical Site #2068, Panorama City, California
  - Viking Clinical Site #2132, Rolling Hills Estates, California
  - Viking Clinical Site #2131, San Diego, California
  - Viking Clinical Site #2052, Spring Valley, California
  - Viking Clinical Site #2109, Tustin, California
  - Viking Clinical Site #2067, Van Nuys, California
  - Viking Clinical Site #2079, Walnut Creek, California
  - Viking Clinical Site #2119, Denver, Colorado
  - Viking Clinical Site #2123, Washington D.C., District of Columbia
  - Viking Clinical Site #2013, Clearwater, Florida
  - Viking Clinical Site #2121, Clearwater, Florida
  - Viking Clinical Site #2003, Cooper City, Florida
  - Viking Clinical Site #2112, DeLand, Florida
  - Viking Clinical Site #2107, Delray Beach, Florida
  - Viking Clinical Site #2083, Fort Myers, Florida
  - Viking Clinical Site #2058, Jacksonville, Florida
  - Viking Clinical Site #2076, Lakeland, Florida
  - Viking Clinical Site #2060, Lakewood Rch, Florida
  - Viking Clinical Site #2117, Miami, Florida
  - Viking Clinical Site #2012, Ocoee, Florida
  - Viking Clinical Site #2056, Palmetto Bay, Florida
  - Viking Clinical Site #2011, Port Orange, Florida
  - Viking Clinical Site #2057, West Palm Beach, Florida
  - Viking Clinical Site #2116, Atlanta, Georgia
  - Viking Clinical Site #2030, Columbus, Georgia
  - Viking Clinical Site #2120, Rincon, Georgia
  - Viking Clinical Site #2093, Savannah, Georgia
  - Viking Clinical Site #2025, Woodstock, Georgia
  - Viking Clinical Site #2062, Honolulu, Hawaii
  - Viking Clinical Site #2080, Meridian, Idaho
  - Viking Clinical Site #2006, Chicago, Illinois
  - Viking Clinical Site #2146, Indianapolis, Indiana
  - Viking Clinical Site #2127, Valparaiso, Indiana
  - Viking Clinical Site #2147, Sioux City, Iowa
  - Viking Clinical Site #2022, West Des Moines, Iowa
  - Viking Clinical Site #2099, Wichita, Kansas
  - Viking Clinical Site #2069, Lexington, Kentucky
  - Viking Clinical Site #2040, Lexington, Kentucky
  - Viking Clinical Site #2009, Louisville, Kentucky
  - Viking Clinical Site #2118, Baton Rouge, Louisiana
  - Viking Clinical Site #2139, Baton Rouge, Louisiana
  - Viking Clinical Site #2106, Lafayette, Louisiana
  - Viking Clinical Site #2020, Metairie, Louisiana
  - Viking Clinical Site #2087, Monroe, Louisiana
  - Viking Clinical Site #2094, Chevy Chase, Maryland
  - Viking Clinical Site #2145, Rockville, Maryland
  - Viking Clinical Site #2066, Rockville, Maryland
  - Viking Clinical Site #2001, Methuen, Massachusetts
  - Viking Clinical Site #2100, Lansing, Michigan
  - Viking Clinical Site #2038, Ypsilanti, Michigan
  - Viking Clinical Site #2140, Gulfport, Mississippi
  - Viking Clinical Site #2031, City of Saint Peters, Missouri
  - Viking Clinical Site #2016, Kansas City, Missouri
  - Viking Clinical Site #2125, Springfield, Missouri
  - Viking Clinical Site #2108, St Louis, Missouri
  - Viking Clinical Site #2010, Butte, Montana
  - Viking Clinical Site #2075, Omaha, Nebraska
  - Viking Clinical Site #2035, Las Vegas, Nevada
  - Viking Clinical Site #2034, Reno, Nevada
  - Viking Clinical Site #2065, Lebanon, New Hampshire
  - Viking Clinical Site #2095, Marlton, New Jersey
  - Viking Clinical Site #2029, Albuquerque, New Mexico
  - Viking Clinical Site #2088, Albany, New York
  - Viking Clinical Site #2042, East Syracuse, New York
  - Viking Clinical Site #2096, Hartsdale, New York
  - Viking Clinical Site #2133, New York, New York
  - Viking Clinical Site #2021, The Bronx, New York
  - Viking Clinical Site #2032, Westfield, New York
  - Viking Clinical Site #2141, Charlotte, North Carolina
  - Viking Clinical Site #2101, Fayetteville, North Carolina
  - Viking Clinical Site #2026, Greensboro, North Carolina
  - Viking Clinical Site #2110, Morehead City, North Carolina
  - Viking Clinical Site #2061, Morehead City, North Carolina
  - Viking Clinical Site #2115, Winston-Salem, North Carolina
  - Viking Clinical Site #2027, Fargo, North Dakota
  - Viking Clinical Site #2043, Cincinnati, Ohio
  - Viking Clinical Site #2074, Cincinnati, Ohio
  - Viking Clinical Site #2044, Cleveland, Ohio
  - Viking Clinical Site #2089, Columbus, Ohio
  - Viking Clinical Site #2148, Dayton, Ohio
  - Viking Clinical Site #2113, Norman, Oklahoma
  - Viking Clinical Site #2137, Tulsa, Oklahoma
  - Viking Clinical Site #2097, Portland, Oregon
  - Viking Clinical Site #2126, Portland, Oregon
  - Viking Clinical Site #2045, East Greenwich, Rhode Island
  - Viking Clinical Site #2028, Greenville, South Carolina
  - Viking Clinical Site #2134, Myrtle Beach, South Carolina
  - Viking Clinical Site #2023, North Charleston, South Carolina
  - Viking Clinical Site #2004, Knoxville, Tennessee
  - Viking Clinical Site #2008, Nashville, Tennessee
  - Viking Clinical Site #2047, Abilene, Texas
  - Viking Clinical Site #2063, Austin, Texas
  - Viking Clinical Site #2007, Austin, Texas
  - Viking Clinical Site #2091, Bellaire, Texas
  - Viking Clinical Site #2124, Brownsville, Texas
  - Viking Clinical Site #2049, Dallas, Texas
  - Viking Clinical Site #2048, Dallas, Texas
  - Viking Clinical Site #2111, Frisco, Texas
  - Viking Clinical Site #2046, Houston, Texas
  - Viking Clinical Site #2077, Lampasas, Texas
  - Viking Clinical Site #2143, San Antonio, Texas
  - Viking Clinical Site #2085, San Antonio, Texas
  - Viking Clinical Site #2015, San Antonio, Texas
  - Viking Clinical Site #2102, Seabrook, Texas
  - Viking Clinical Site #2002, Ogden, Utah
  - Viking Clinical Site #2092, Salt Lake City, Utah
  - Viking Clinical Site #2039, Sandy City, Utah
  - Viking Clinical Site #2024, St. George, Utah
  - Viking Clinical Site #2098, Arlington, Virginia
  - Viking Clinical Site #2082, Suffolk, Virginia
  - Viking Clinical Site #2072, Renton, Washington
  - Viking Clinical Site #2041, Spokane, Washington
- Puerto Rico (2):
  - Viking Clinical Site #2130, Mayagüez
  - Viking Clinical Site #2086, San Juan